CLINICAL TRIAL: NCT04162600
Title: A Phase I Clinical Trial to Determine the Safety and Immunogenicity of the Candidate Rabies Vaccine ChAdOx2 RabG in UK Healthy Adult Volunteer
Brief Title: Safety and Immunogenicity of the Candidate Rabies Vaccine ChAdOx2 RabG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Since acceptable safety, tolerability, and immunogenicity was demonstrated at the highest dose tested (group 3, fully recruited), there was no scientific or ethical justification to recruit more participants into the mid-dose group (group 2).
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAB001
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-07

CONDITIONS: Rabies
Keywords: Vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5 x 10^9 vp of ChAdOx2 RabG (Experimental): Volunteers will receive a standalone dose of ChAdOx2 RabG 5 x 10^9 vp vaccination intramuscularly. Optional extended follow-up, volunteers will receive a complete pre-exposure prophylactic course of an existing rabies vaccine.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- 2.5 x 10^10 vp of ChAdOx2 RabG (Experimental): Volunteers will receive a standalone dose of ChAdOx2 RabG 2.5 x 10^10 vp vaccination intramuscularly. Optional extended follow-up, volunteers will receive a complete pre-exposure prophylactic course of an existing rabies vaccine.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine
- 5 x 10^10 vp of ChAdOx2 RabG (Experimental): Volunteers will receive a standalone dose of ChAdOx2 RabG 5 x 10^10 vp vaccination intramuscularly. Optional extended follow-up, volunteers will receive a complete pre-exposure prophylactic course of an existing rabies vaccine.
  Interventions: Biological: ChAdOx2 RabG; Biological: Inactivated Rabies Vaccine

INTERVENTIONS:
Biological: ChAdOx2 RabG — Single dose of ChAdOx2 RabG at different concentrations: 5 x 10^9 vp, 2.5 x 10^10 vp, 5 x 10^10 vp
  Arms: 2.5 x 10^10 vp of ChAdOx2 RabG
Biological: Inactivated Rabies Vaccine — A complete pre-exposure prophylactic course of an existing rabies vaccine, ≥2.5 international units.
  Arms: 2.5 x 10^10 vp of ChAdOx2 RabG
Biological: ChAdOx2 RabG — Single dose of ChAdOx2 RabG at different concentrations: 5 x 10^9 vp, 2.5 x 10^10 vp, 5 x 10^10 vp
  Arms: 5 x 10^10 vp of ChAdOx2 RabG
Biological: ChAdOx2 RabG — Single dose of ChAdOx2 RabG at different concentrations: 5 x 10^9 vp, 2.5 x 10^10 vp, 5 x 10^10 vp.
  Arms: 5 x 10^9 vp of ChAdOx2 RabG
Biological: Inactivated Rabies Vaccine — A complete pre-exposure prophylactic course of an existing rabies vaccine, ≥2.5 international units.
  Arms: 5 x 10^10 vp of ChAdOx2 RabG
Biological: Inactivated Rabies Vaccine — A complete pre-exposure prophylactic course of an existing rabies vaccine, ≥2.5 international units.
  Arms: 5 x 10^9 vp of ChAdOx2 RabG

SUMMARY:
This is a first-in-human, open-label, dose escalation, phase I clinical trial to assess the safety and immunogenicity of the candidate ChAdOx2 RabG vaccine in healthy UK volunteers aged 18-65. The vaccine will be administered intramuscularly (IM).

DETAILED DESCRIPTION:
Volunteers will be recruited and vaccinated at the Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Oxford. There will be 3 study groups and it is anticipated that a total of 12 volunteers will be enrolled. Staggered enrolment will apply between study groups and for the first three volunteers within each group.

The study includes an optional extended follow-up period, lasting one month and starting one year after vaccination. Volunteers will receive a complete pre-exposure prophylactic course of an existing rabies vaccine, allowing study of the immunological memory (recall response) induced by ChAdOx2 RabG. A second optional element of the study is the collection of saliva samples at each visit for the study of shedding of EBV and CMV.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 65 years.
2. Able and willing (in the Investigator's opinion) to comply with all study requirements.
3. Willing to allow the investigators to discuss the volunteer's medical history with their GP.
4. For females only, willingness to practice continuous effective contraception during the study and a negative pregnancy test on the day(s) of screening and vaccination(s).
5. Agreement to refrain from blood donation during the course of the study.
6. Provide written informed consent.

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period. To be re- confirmed at the enrolment visit.
2. Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data (e.g. Adenovirus vectored vaccine).
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
6. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
7. Any history of anaphylaxis in relation to vaccination.
8. Pregnancy, lactation or willingness/intention to become pregnant during the study.
9. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
10. History of serious psychiatric condition likely to affect participation in the study.
11. Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture.

13. Individuals who have previously experienced episodes of capillary leak syndrome.

14. History of confirmed major thrombotic event (including cerebral venous sinus thrombosis, deep vein thrombosis, pulmonary embolism).

15. History of antiphospholipid syndrome. 16. History of prior receipt of unfractionated heparin. 17. History of heparin induced thrombocytopenia. 18. Any other serious chronic illness requiring hospital specialist supervision.

19. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week. 20. Suspected or known injecting drug abuse in the 5 years preceding enrolment. 21. Detectable circulating hepatitis B surface antigen (HBsAg). 22. Seropositive for hepatitis C virus (antibodies to HCV). 23. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis. 24. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.

25. Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate. 26. Receipt of any prior rabies vaccine, including an incomplete course. 27. Require or will require rabies vaccination during the first 8 weeks of the study period (e.g. through planned travel to high risk enzootic areas of through work which may lead to exposure and for which rabies vaccination is usually required/recommended).

Exclusion criteria for optional follow-up

1. Receiving rabies vaccination following the completion of the first 8 weeks of follow-up but before the optional extended follow-up period will exclude participants from taking part in the optional follow-up period.
2. History of allergic reactions to amphotericin B, chlortetracycline, neomycin, polymyxin, streptomycin, or to any antibiotics of the same groups will exclude participants from receiving certain IRVs (as per the relevant SmPC) during the optional extended follow-up period, but will not exclude participants from receiving ChAdOx2 RabG.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ChAdOx2 RabG in healthy volunteers given as a standalone vaccine at different doses assessed by the occurrence of solicited adverse events. | Assessment of solicited AEs in the first 7 days post vaccination
  Occurrence of solicited local and systemic adverse events (i.e: pain, redness, swelling and pruritus at injection site and temperature, feverishness, myalgia, arthralgia, malaise, headache, fatigue and nausea).
Safety and tolerability of ChAdOx2 RabG in healthy volunteers given as a standalone vaccine at different doses assessed by the occurrence of solicited adverse events. | Unsolicited AEs to be assessed up to 28 days post vaccination.
  Occurrence of unsolicited local and systemic adverse events
Safety and tolerability of ChAdOx2 RabG in healthy volunteers given as a standalone vaccine at different doses assessed by the occurrence of serious adverse events. | SAEs will be collected from enrolment until the end of the follow-up period.(8 weeks)
  Occurrence of serious adverse events
Safety and tolerability of ChAdOx2 RabG in healthy volunteers given as a standalone vaccine at different doses assessed by the occurrence of solicited adverse events. | At Day 0 (baseline), day 2, day 7, day 28 and day 56 post vaccination
  Occurrence of laboratory adverse events defined as clinically significant changes from baseline. Haematology (Full Blood Count) and Biochemistry (Kidney and Liver Function Tests) will be assessed.

SECONDARY OUTCOMES:
Immunogenicity of the ChAdOx2 RabG vaccine | Day 365
  Rapid fluorescent focus inhibition test (RFFIT) of virus neutralising antibody

OTHER OUTCOMES:
Immunological memory induced by ChAdOx2 RabG | Between days 365 and 386
  Virus neutralizing antibody will be measured before and in the course of immunisation with IRVs during an optional extended follow-up.
Timecourse of EBV and CMV shedding | Study Duration (386 days)
  Measured by quantitative PCR.
Level of EBV and CMV shedding | Study Duration (386 days)
  Measured by quantitative PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Douglas, Principal Investigator — Jenner Institute
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

REFERENCES:
- [Derived] Jenkin D, Ritchie AJ, Aboagye J, Fedosyuk S, Thorley L, Provstgaad-Morys S, Sanders H, Bellamy D, Makinson R, Xiang ZQ, Bolam E, Tarrant R, Ramos Lopez F, Platt A, Poulton I, Green C, Ertl HCJ, Ewer KJ, Douglas AD. Safety and immunogenicity of a simian-adenovirus-vectored rabies vaccine: an open-label, non-randomised, dose-escalation, first-in-human, single-centre, phase 1 clinical trial. Lancet Microbe. 2022 Sep;3(9):e663-e671. doi: 10.1016/S2666-5247(22)00126-4. Epub 2022 Jul 27. PMID 35907430